CLINICAL TRIAL: NCT02392247
Title: Hemosonics- VCU Cardiac Surgery Clinical Study Protocol
Brief Title: Hemosonics- VCU Cardiac Surgery Clinical Study
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: HemoSonics LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: FTU-002-007
Record Dates: First submitted 2015-03-12; First posted 2015-03-18 (Estimated); Results first posted 2016-07-12 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-06

CONDITIONS: Cardiopulmonary Bypass

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiac Surgery Patients: Single cohort of 50 consecutive cardiac surgery patients undergoing cardiopulmonary bypass. The study compares output of two technologies for determination of point of care coagulation function: thromboelastography (TEG; current care option) and the new technology Sonic Estimation of Elasticity via Resonance (SEER) Sonorheometry
  Interventions: Device: Coagulation function

INTERVENTIONS:
Device: Coagulation function — Coagulation function assessment tools TEG (standard of practice) vs SEER Quantra (novel coagulation function device)

SUMMARY:
This study compares the results of current standard coagulation measurement devices to the Quantra System, a new device, using small amount of extra blood obtained during routine blood draws in cardiac surgery patients.

DETAILED DESCRIPTION:
HemoSonics is developing a novel POC diagnostic device, the Quantra System, to perform whole blood coagulation analysis and which is suitable for use in surgical and intensive care settings. The Quantra System employs a patented technology named sonorheometry, which was invented at the University of Virginia. Sonorheometry uses ultrasound pulses to characterize the dynamic changes in viscoelastic properties of a blood sample during coagulation and clot lysis. The initial assay performed on the Quantra System will be the surgical assay for monitoring hemostasis during major surgical procedures in adult patients.

A clinical study will be conducted to evaluate the analytical performance as well as provide a preliminary evaluation of the performance comparability of the HemoSonics' device as compared to existing coagulation monitoring technology in heart surgery. This study will be performed at HemoSonics and the Virginia Commonwealth University Medical Center and will involve patients undergoing cardiac surgery requiring bypass.

ELIGIBILITY:
Inclusion Criteria:

* Subject is scheduled for cardiac surgery involving bypass circuit
* Subject is older than 18 years
* Subject is willing to participate and he/she has signed a consent form

Exclusion Criteria:

* Subject is unable to provide written informed consent
* Subject is incarcerated at the time of the study
* Subject is affected by any condition that, in the opinion of the surgical team, may pose additional risks
* Patients on emergency cases

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants for this study will be recruited at the Virginia Commonwealth University Medical Center. The subject population will be representative of the local racial and ethnic population.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2015-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Speiss, M.D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cardiac Surgery Patients: Single cohort of 50 consecutive cardiac surgery patients undergoing cardiopulmonary bypass. The study compares output of two technologies for determination of point of care coagulation function: thromboelastography (TEG; current care option) and the new technology Sonic Estimation of Elasticity via Resonance (SEER) Sonorheometry. Blood was collected at four time points: baseline, during bypass, 10 minutes after heparin reversal just prior to bypass weaning, and off-bypass before transfer to the ICU.
  Blood specimen collection
Period: Overall Study
Arm/Group | Cardiac Surgery Patients
Started | 52
Completed | 50
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Surgery cancelled; no data | 1

BASELINE CHARACTERISTICS:
Groups:
- Cardiac Surgery Patients: Single cohort of 50 consecutive cardiac surgery patients undergoing cardiopulmonary bypass. Paired blood samples were assessed by thromboelastography (TEG; current care option) and by Sonic Estimation of Elasticity via Resonance (SEER) Sonorheometry
Arm/Group | Cardiac Surgery Patients
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 33
  >=65 years | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 17
  White | 27
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Clot Time
Description: Coagulation Function assessed at 4 time points [baseline, during bypass, 10 minutes after heparin reversal just prior to bypass weaning, and off-bypass before transfer to the ICU] over the course of cardiac surgery until patient ICU transfer
Time Frame: 1 day
Population: Matched paired blood samples evaluating coagulation function by two methods (TEG, SEER) obtained from each patient at each sampling time (baseline, during bypass, 10 minutes after heparin reversal just prior to bypass weaning, and off-bypass before transfer to the ICU)
Measure: Mean (Standard Deviation); unit: min
Units Other Than Participants: blood samples
Arm/Group | Cardiac Surgery Patients
Number analyzed (Participants) | 50
Number analyzed (blood samples) | 200
min
  Reaction Time R (TEG) | 4.9 (1.2)
  Heparinase Clot Time (SEER) | 3.3 (0.6)
Statistical Analysis 1: Comparison: Cardiac Surgery Patients; A cohort of 50 patients was estimated to capture at least 7 'bleeding' patients with a likelihood of 95%, assuming a 25% incidence of bleeding, and standard deviation of 20%, to determine maximum clot stiffness within +/- 10% of the mean. This was a descriptive and method-comparison study. Method comparisons were performed according to Clinical Laboratory Science Institute (CLSI) guidelines (Deming regression on paired measurements); Test type: Superiority or Other; p < 0.001, Deming Regression — This study was not designed to determine which method is 'superior'.Statistical significance refers to deviation of slope for perfect agreement (=1) between paired measurements to quantify strength of association; Slope = 0.34, 95% CI 2-sided [0.26 to 0.44] — Slope measured deviation from 1:1 concordance between SEER and TEG with TEG measurement as denominator. Confidence intervals were obtained by bootstrapping 1000 times on the parameters estimates for the slopes, intervals and correlation coefficients

2. Primary Outcome: Clot Stiffness
Description: Coagulation Function assessed at 4 time points (baseline, during bypass, 10 minutes after heparin reversal just prior to bypass weaning, and off-bypass before transfer to the ICU) over the course of cardiac surgery and bypass until patient ICU transfer
Time Frame: 1 day
Population: Matched paired blood samples evaluating coagulation function by two methods (TEG, SEER) for each patient at each of 4 time points [baseline, during bypass, 10 minutes after heparin reversal just prior to bypass weaning, and off-bypass before transfer to the ICU]
Measure: Mean (Standard Deviation); unit: hPa
Units Other Than Participants: blood samples
Arm/Group | Cardiac Surgery Patients
Number analyzed (Participants) | 50
Number analyzed (blood samples) | 200
hPa
  TEG G force | 8.5 (3.7)
  SEER Clot stiffness | 18.4 (9.2)
Statistical Analysis 1: Comparison: Cardiac Surgery Patients; A cohort of 50 patients was estimated to capture at least 7 'bleeding' patients with a likelihood of 95%, assuming a 25% incidence of bleeding, and standard deviation of 20%, to determine maximum clot stiffness within +/- 10% of the mean. This was a descriptive and method-comparison study. Method comparisons were performed according to Clinical Laboratory Science Institute (CLSI) guidelines (Deming regression on paired measurements ); Test type: Superiority or Other; p < 0.001, Deming regression — This study was not designed to determine which method is 'superior'. Statistical significance refers to deviation of slope for perfect agreement (=1) between paired measurements to quantify strength of association; Confidence intervals were obtained by bootstrapping 1000 times on the parameters estimates for the slopes, intervals and correlation coefficients; Slope = 3.1, 95% CI 2-sided [2.9 to 3.4] — Slope measured deviation from 1:1 concordance between SEER and TEG with TEG as denominator. Confidence intervals were obtained by bootstrapping 1000 times on the parameters estimates for the slopes, intervals and correlation coefficients

ADVERSE EVENTS:
Time Frame: one day
Description: 'Bleeding' was defined as chest tube drainage > 1500 mL in 24 hr; serious bleeding was defined as necessitating a return to the operating room for re-exploration.
Groups:
- Cardiac Surgery Patients: Single cohort of 50 consecutive cardiac surgery patients undergoing cardiopulmonary bypass. The study compares output of two technologies for determination of point of care coagulation function: thromboelastography (TEG; current care option) and the new technology Sonic Estimation of Elasticity via Resonance (SEER) Sonorheometry
  Blood specimen collection
Arm/Group | Cardiac Surgery Patients
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

LIMITATIONS AND CAVEATS:
This is a descriptive, single-cohort study, not an hypothesis-testing trial. The objective was device performance comparison. As there is no gold standard technology, this study could not determine which method was 'best' or 'superior'.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No